CLINICAL TRIAL: NCT04445831
Title: A Phase Ib/IIa Multicenter, Double-Blind, Randomized, Placebo-Controlled Study to Evaluate the Safety, Tolerability and Immunogenicity of Different Doses, Regimens and Combinations of Tau Targeted Vaccines in Subjects With Early Alzheimer's Disease
Brief Title: A Study to Evaluate the Safety, Tolerability and Immunogenicity of Tau Targeted Vaccines in Participants With Early Alzheimer's Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AC Immune SA (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACI-35-1802; 2018-004573-27 (EudraCT Number)
Record Dates: First submitted 2020-06-22; First posted 2020-06-24 (Actual); Results first posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-01

CONDITIONS: Alzheimer's Disease; Cognitive Impairment; Tauopathies; Mild Cognitive Impairment; Dementia; Brain Diseases; Central Nervous System Diseases
Keywords: Alzheimer's Disease; Cognitive Impairment; Tauopathies; Mild Cognitive Impairment; Dementia; Brain Diseases; Central Nervous System Diseases
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Tauopathies; Dementia; Brain Diseases; Central Nervous System Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Placebo (Placebo Comparator): Placebo administered at predefined time points over a 48-week period.
  Interventions: Other: Placebo
- ACI-35.030 - Low dose (Experimental): Active vaccine administered at predefined time points over a 48-week period.
  Interventions: Biological: ACI-35.030
- ACI-35.030 - Medium dose (Experimental): Active vaccine administered at predefined time points over a 48-week period.
  Interventions: Biological: ACI-35.030
- ACI-35.030 - High dose (Experimental): Active vaccine administered at predefined time points over a 48-week period.
  Interventions: Biological: ACI-35.030
- JACI-35.054 - Low dose (Experimental): Active vaccine administered at predefined time points over a 48-week period.
  Interventions: Biological: JACI-35.054
- JACI-35.054 - Medium dose (Experimental): Active vaccine administered at predefined time points over a 48-week period.
  Interventions: Biological: JACI-35.054

INTERVENTIONS:
Biological: ACI-35.030 — Administration of a Low dose of ACI-35.030
  Arms: ACI-35.030 - Low dose
Biological: ACI-35.030 — Administration of a Medium dose of ACI-35.030
  Arms: ACI-35.030 - Medium dose
Biological: ACI-35.030 — Administration of a High dose of ACI-35.030
  Arms: ACI-35.030 - High dose
Other: Placebo — Administration of Placebo
  Arms: Placebo
Biological: JACI-35.054 — Administration of a Low dose of JACI-35.054
  Arms: JACI-35.054 - Low dose
Biological: JACI-35.054 — Administration of a Medium dose of JACI-35.054
  Arms: JACI-35.054 - Medium dose

SUMMARY:
This study is a multicenter, double blind, randomized, placebo-controlled study to evaluate the safety, tolerability and immunogenicity of different doses, regimens and combinations of Tau targeted vaccines in participants with early Alzheimer's Disease.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female with age from 50 and up to 75 years old inclusive.
2. Mild Cognitive Impairment (MCI) due to AD or Mild AD according to NIA-AA criteria and Clinical Dementia Rating scale (CDR) global score of 0.5 or 1 respectively.
3. Mini Mental State Examination (MMSE) score of 22 or above.
4. Abnormal level of CSF Abeta amyloid 42 (Aß42) consistent with AD pathology at screening.
5. Subjects either not taking any marketed treatment for AD or receiving a stable dose of an acetylcholinesterase inhibitor and/or memantine for at least 3 months prior to baseline.
6. Subjects cared for by a reliable informant or caregiver to assure compliance, assist with clinical assessments and report safety issues.
7. Women must be post-menopausal for at least one year and/or surgically sterilized.
8. Subjects who in the opinion of the investigator is able to understand and provide written informed consent.
9. Both subject and informant or caregiver must be fluent in one of the languages of the study and able to comply with all study procedures, including lumbar punctures.

Exclusion criteria:

1. Participation in previous clinical trials for AD and/or for neurological disorders using active immunization unless there is documented evidence that the subject was treated with placebo only and the placebo vaccine is not expected to induce any specific immune response.
2. Participation in previous clinical trials for AD and/or for neurological disorders using any passive immunization within the past 6 months (or 5 half-lives of the investigational antibody, whichever is longer) prior to screening unless there is documented evidence that the subject was treated with placebo only and the placebo is not expected to induce any specific immune response.
3. Participation in previous clinical trials for AD and/or for neurological disorders using any small molecule drug including BACE-1 inhibitors within the past 3 months prior to screening.
4. Concomitant participation in any other clinical trial using experimental or approved medications or therapies.
5. Presence of positive Anti-nuclear Antibody (ANA) titers at a dilution of at least 1:160 in subjects without clinical symptoms of auto-immune disease.
6. Current or past history of auto-immune disease, or clinical symptoms consistent with the presence of auto-immune disease.
7. Immune suppression including but not limited to the use of immunosuppressive drugs or systemic steroids unless they have been prescribed transiently more than 3 months prior to screening.
8. History of severe allergic reaction (e.g., anaphylaxis) including but not limited to severe allergic reaction to previous vaccines and/or medications.
9. Prior history of clinically significant hypoglycaemic episodes.
10. Drug or alcohol abuse or dependence currently met or within the past five years according to Diagnostic and Statistical Manual of Mental Disorders-V (DSM-V) criteria.
11. Any clinically significant medical condition likely to interfere with the evaluation of safety and tolerability of the study treatment and/or the adherence to the full study visit schedule.
12. Any clinically significant medical condition likely to impact the immune system (e.g, any history of acquired or innate immune system disorder).
13. Use of hydralazine, procainamide, quinidine, isoniazide, TNF-inhibitors, minocycline within the last 12 months prior to screening.
14. Use of diltiazem unless on a stable dose for at least 3 months prior to screening.
15. Significant risk of suicide defined, using the Columbia-Suicide Severity Rating Scale, as the subject answering: "yes" to suicidal ideation questions 4 or 5 or answering: "yes" to suicidal behavior within the past 12 months.
16. Concomitant psychiatric or neurologic disorder other than those considered to be related to AD.
17. History or presence of uncontrolled seizures.
18. History of meningoencephalitis within the past 10 years prior to screening.
19. Subjects with a history of hemorrhagic and/or non-hemorrhagic stroke.
20. Presence or history of peripheral neuropathy.
21. History of inflammatory neurological disorders with potential for CNS involvement.
22. Screening MRI scan showing structural evidence of alternative pathology not consistent with AD which could cause the subject's symptoms.
23. MRI examination cannot be done for any reason, including but not limited to metal implants contraindicated for MRI studies and/or severe claustrophobia.
24. Significant hearing or visual impairment or other issues judged relevant by the investigator preventing to comply with the protocol and to perform the outcome measures.
25. Clinically significant infections or major surgical operation within 3 months prior to screening.
26. Any vaccine received within the past 2 weeks before screening, including influenza vaccine.
27. Clinically significant arrhythmias or other clinically significant abnormalities on ECG at screening.
28. Myocardial infarction within one year prior to baseline, unstable angina pectoris, or significant coronary artery disease.
29. History of cancer within the past 5 years other than treated squamous cell carcinoma, basal cell carcinoma and melanoma in situ, or in-situ prostate cancer or in-situ breast cancer which have been fully removed and are considered cured.
30. Clinically significant deviations from normal values for hematologic parameters, liver function tests, and other biochemical measures, that are judged to be clinically significant in the opinion of the investigator.
31. Pregnancy confirmed by blood test at screening, or subject planning to be pregnant or lactating.
32. Receipt of any anticoagulant drug or antiplatelet drug, except aspirin at doses of 100 mg daily or lower.
33. Receipt of any antipsychotic drugs unless on stable low doses for the treatment of insomnia.
34. Donation of blood or blood products within 30 days prior to screening or plans to donate blood while participating in the study.
35. Positive Venereal Disease Research Laboratory (VDRL) consistent with active syphilis at screening.
36. Positive HIV test at screening.
37. Laboratory or clinical evidence of active hepatitis B and/or C at screening.
38. Serum creatinine greater than 1.5x upper limit of normal, abnormal thyroid function tests or clinically significant reduction in serum B12 or folate levels.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2019-07-31 (Actual); Primary Completion 2023-09-05 (Actual); Study Completion 2023-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Scheltens, MD, Principal Investigator — Amsterdam UMC Alzheimer Center de Boelelaan Amsterdam The Netherlands
Locations (9):
- Finland (3):
  - Clinical Research Services Helsinki, Helsinki
  - Itä-Suomen Yliopisto - Kuopion Kampus, Kuopio
  - Clinical Research Services Turku, Turku
- Netherlands (2):
  - Brain Research Center - Den Bosch, 's-Hertogenbosch
  - Brain Research Center - Amsterdam, Amsterdam
- Sweden (2):
  - Minnesmottagningen - Sahlgrenska Universitetssjukhuset - Mölndal Sjukhus, Mölndal
  - Kognitiv Mottagning - Karolinska Universitetssjukhuset - Huddinge, Stockholm
- United Kingdom (2):
  - Edinburgh Clinical Research Facility, Edinburgh
  - University College London Hospitals NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) are not planned to be shared for this early-phase non-pivotal ACI-35-1802 Phase 1b/2a study. However, group-level data may be shared to qualified researchers who engage in rigorous independent scientific research after the review and approval of a proposal sent to the sponsor (see Contacts) and the execution of a data sharing agreement.
  In addition, the Clinical Study Protocol and the Statistical Plan will be available in this registry once the study results are released.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was performed in Finland, the Netherlands, Sweden and the UK. 79 subjects were screened for the study; 22 subjects did not meet the eligibility criteria; 1 subject was re-screened and qualified to participate.
Pre-assignment Details: Screening details:
  Subjects between 50 and 75 years at screening with Mild Cognitive Impairment (MCI) due to AD or Mild AD according to NIA-AA criteria, providing a written informed consent and fulfilling all further inclusion criteria could enter the clinical trial.
Groups:
- Sub-Cohort 1.1 (ACI-35.030 300 μg): Subjects receiving 4 doses of ACI-35.030 300 μg at week 0, 8, 24 and 48
- Sub-Cohort 1.2 (ACI-35.030 900 μg): Subjects receiving 4 doses of ACI-35.030 900 μg at week 0, 8, 24 and 48
- Sub-Cohort 1.3 (ACI-35.030 1800 μg): Subjects receiving 4 doses of ACI-35.030 1800 μg at week 0, 8, 24 and 48
- Cohort 1 Placebo: Subjects receiving 4 doses of placebo at week 0, 8, 24 and 48. The placebo subjects of the 3 sub-cohorts 1.1, 1.2 and 1.3 (cohort 1) are pooled to represent one group. Randomization and distribution of the subjects in cohort 1 was as follows:
  * Cohort 1.1: 8 patients (6 active, 2 placebo)
  * Cohort 1.2: 25 patients (19 active, 6 placebo)
  * Cohort 1.3: 8 patients (6 active, 2 placebo)
- Sub-Cohort 2.1 (JACI-35.054 15 μg): Subjects receiving 4 doses of JACI-35.054 15 μg at week 0, 8, 24 and 48
- Sub-Cohort 2.2 (JACI-35.054 60 μg): Subjects receiving 4 doses of JACI-35.054 60 μg at week 0, 8, 24 and 48
- Cohort 2 Placebo: Subjects receiving 4 doses of placebo at week 0, 8, 24 and 48. The placebo subjects of the 2 sub cohorts 2.1 and 2.2 (cohort 2) are pooled to represent one group. Randomization and distribution of the subjects in cohort 2 was as follows:
  * Cohort 2.1: 8 patients (6 active, 2 placebo)
  * Cohort 2.2: 8 patients (6 active, 2 placebo)
Period: Overall Study
Arm/Group | Sub-Cohort 1.1 (ACI-35.030 300 μg) | Sub-Cohort 1.2 (ACI-35.030 900 μg) | Sub-Cohort 1.3 (ACI-35.030 1800 μg) | Cohort 1 Placebo | Sub-Cohort 2.1 (JACI-35.054 15 μg) | Sub-Cohort 2.2 (JACI-35.054 60 μg) | Cohort 2 Placebo
Started | 6 | 19 | 6 | 10 | 6 | 6 | 4
Completed | 4 | 17 | 5 | 10 | 6 | 6 | 4
Not Completed | 2 | 2 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Subject withdrawal by caregiver | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The data of the 57 subjects who have been randomized in the study (e.g. signed the consent, eligible and received at east 1 administration of the study drug) have been considered
Groups:
- Total: Total of all reporting groups
Arm/Group | Sub-Cohort 1.1 (ACI-35.030 300 μg) | Sub-Cohort 1.2 (ACI-35.030 900 μg) | Sub-Cohort 1.3 (ACI-35.030 1800 μg) | Cohort 1 Placebo | Sub-Cohort 2.1 (JACI-35.054 15 μg) | Sub-Cohort 2.2 (JACI-35.054 60 μg) | Cohort 2 Placebo | Total
Number analyzed (Participants) | 6 | 19 | 6 | 10 | 6 | 6 | 4 | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 6 | 2 | 2 | 1 | 5 | 1 | 20
  >=65 years | 3 | 13 | 4 | 8 | 5 | 1 | 3 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.5 (5.01) | 68.0 (6.29) | 64.7 (4.63) | 67.7 (4.60) | 66.7 (6.22) | 63.0 (4.77) | 68.0 (6.16) | 66.67 (5.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 9 | 2 | 5 | 3 | 3 | 4 | 30
  Male | 2 | 10 | 4 | 5 | 3 | 3 | 0 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 18 | 6 | 10 | 6 | 6 | 4 | 56
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 6 | 19 | 6 | 10 | 6 | 6 | 4 | 57
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Netherlands | 0 | 6 | 2 | 2 | 3 | 1 | 0 | 14
  Sweden | 0 | 4 | 0 | 1 | 0 | 1 | 0 | 6
  Finland | 6 | 6 | 2 | 7 | 3 | 4 | 4 | 32
  United Kingdom | 0 | 3 | 2 | 0 | 0 | 0 | 0 | 5
Clinical Dementia Rating (CDR) - Global Score [Count of Participants; unit: Participants] — The CDR Scale is used to assess the function of AD subjects in six categories: memory, orientation, judgement and problem solving, community affairs, home and hobbies and personal care. It is based on an interview of the subject and caregiver. Each category is scored from 0 (no symptoms) to 3 (severe). The CDR global score is derived from scores of each individual category (obtained after computation with an algorithm) and ranges from 0 to 3 (severity of symptoms: 0=normal, 0.5 = very mild, 1=mild, 2=moderate, 3=severe). This score was an inclusion criteria (score of 0.5 or 1 at Screening).
  Participants
    Score = 0.5 | 6 | 17 | 5 | 8 | 6 | 5 | 3 | 50
    Score = 1 | 0 | 2 | 1 | 2 | 0 | 1 | 1 | 7
Concomitant Medication [Count of Participants; unit: Participants] — Number of subjects under Acetylcholinesterase Inhibitors and/or Memantine medication at baseline (prior to first dosing).
  Participants
    Acetylcholinesterase Inhibitors and/or Memantine | 5 | 14 | 5 | 8 | 3 | 5 | 4 | 44
    No Acetylcholinesterase Inhibitors or Memantine | 1 | 5 | 1 | 2 | 3 | 1 | 0 | 13
Mini Mental State Examination (MMSE) Total score [Mean (Standard Deviation); unit: units on a scale] — The Mini Mental State Examination (MMSE) is a widely used test of overall cognitive function, assessing memory, orientation and praxis in a short series of tests and questions. The total score (sum of score for each test question) ranges from 0 to 30 with 30 being the best possible score and 0 being the worst possible score. This score was part of the inclusion criteria (score of 22 or above at Screening).
  units on a scale | 27.5 (0.84) | 26.1 (2.02) | 26.0 (2.68) | 26.1 (3.11) | 28.0 (1.55) | 25.7 (3.61) | 24.5 (2.52) | 26.28 (2.46)

OUTCOME MEASURES:

1. Primary Outcome: Overview of Treatment-Emergent Adverse Events, Safety Set
Description: Categorical data are presented with the number of subjects with at least one event for the defined categories. Subjects are included only once, even if they experienced multiple events in a category.
Time Frame: AEs falling between first dosing (week 0) and last study visit (week 74), ie up to 74 weeks, defined as Treatment-Emergent Adverse Events (TEAEs)
Population: Observations are given for the Safety population (all randomized subjects who received at least one dose of the study drug, analyzed based on the study treatment actually received). All 57 subjects randomized in the study received at least 1 dose of the study drug according to their randomized treatment and are therefore all included in the Safety population, which is identical to the Intention-to Treat (ITT) population (all randomized subjects who received at least one dose of the study drug).
Measure: Count of Participants; unit: Participants
Arm/Group | Sub-Cohort 1.1 (ACI-35.030 300 μg) | Sub-Cohort 1.2 (ACI-35.030 900 μg) | Sub-Cohort 1.3 (ACI-35.030 1800 μg) | Cohort 1 Placebo | Sub-Cohort 2.1 (JACI-35.054 15 μg) | Sub-Cohort 2.2 (JACI-35.054 60 μg) | Cohort 2 Placebo
Number analyzed (Participants) | 6 | 19 | 6 | 10 | 6 | 6 | 4
Participants
  Any TEAE | 6 | 17 | 6 | 8 | 6 | 6 | 4
  Any Serious TEAE | 2 | 2 | 2 | 0 | 0 | 0 | 1
  Any Severe TEAE | 1 | 2 | 0 | 0 | 0 | 0 | 1
  Any Adverse Drug Reactions | 3 | 15 | 6 | 2 | 4 | 2 | 0
  Any Serious Adverse Drug Reactions | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Any TEAE Leading to Study Drug Discontinuation | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any TEAE Leading to Study Discontinuation | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any TEAE with Outcome of Death | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Overview of Treatment-Emergent Adverse Events Assessed by Intensity, Safety Set
Description: Categorical data are presented with the number of subjects with at least one Treatment-Emergent Adverse Event (TEAE) assessed as:
  * Mild: Easily tolerated and causes minimal discomfort and does not interfere with everyday activities.
  * Moderate: Sufficiently discomforting to interfere with normal everyday activities; intervention may be needed. Event is not hazardous to the subject's health
  * Severe: Prevents normal everyday activities; treatment or other intervention usually needed. Hazard to the subject's health
  Although subjects may have experienced multiple events, they are included only once, in the maximum severity category
Time Frame: Between the first dosing and the last study visit (week 74)
Population: Observations are given for the Safety population (all randomized subjects who received at least one dose of the study drug, analyzed based on the study treatment actually received). All 57 subjects randomized in the study received at least 1 dose of the study drug according to their randomized treatment and are therefore all included.
Measure: Count of Participants; unit: Participants
Arm/Group | Sub-Cohort 1.1 (ACI-35.030 300 μg) | Sub-Cohort 1.2 (ACI-35.030 900 μg) | Sub-Cohort 1.3 (ACI-35.030 1800 μg) | Cohort 1 Placebo | Sub-Cohort 2.1 (JACI-35.054 15 μg) | Sub-Cohort 2.2 (JACI-35.054 60 μg) | Cohort 2 Placebo
Number analyzed (Participants) | 6 | 19 | 6 | 10 | 6 | 6 | 4
Participants
  Mild | 2 | 8 | 3 | 4 | 3 | 1 | 2
  Moderate | 3 | 7 | 3 | 4 | 3 | 5 | 1
  Severe | 1 | 2 | 0 | 0 | 0 | 0 | 1

3. Primary Outcome: Overview of Treatment-Emergent Adverse Events Assessed by Relationship to Study Drug, Safety Set
Description: Categorical data are presented with the number of subjects with at least one Treatment-Emergent Adverse Event (TEAE) assessed as:
  * Unrelated: Events reported as unrelated or unlikely related to study drug
  * Related: Events reported as possibly related or probably related to study drug
  Although subjects may have experienced multiple events, they are included only once, in the strongest relationship category
Time Frame: Between the first dosing and the last study visit (week 74)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Sub-Cohort 1.1 (ACI-35.030 300 μg) | Sub-Cohort 1.2 (ACI-35.030 900 μg) | Sub-Cohort 1.3 (ACI-35.030 1800 μg) | Cohort 1 Placebo | Sub-Cohort 2.1 (JACI-35.054 15 μg) | Sub-Cohort 2.2 (JACI-35.054 60 μg) | Cohort 2 Placebo
Number analyzed (Participants) | 6 | 19 | 6 | 10 | 6 | 6 | 4
Participants
  Unrelated | 3 | 2 | 0 | 6 | 2 | 4 | 4
  Related | 3 | 15 | 6 | 2 | 4 | 2 | 0

4. Primary Outcome: Mean Change From Baseline in Diastolic Blood Pressure, ITT Set
Description: At reported visits, diastolic blood pressures (mmHg = millimeter of mercury) were measured in sitting position only, after the subject has been sitting down for at least 5 minutes.
  A change from baseline value is defined as the value at post-baseline timepoint minus the baseline value, i.e. post-baseline value - baseline value
Time Frame: Endpoint is assessed from baseline (i.e. last non-missing value prior to the first immunization at week 0) to the last study visit (week 74), at weeks 26, 50 and 74.
Population: ITT population (i.e. all randomized subjects who received at least 1 dose of the study drug).
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Sub-Cohort 1.1 (ACI-35.030 300 μg) | Sub-Cohort 1.2 (ACI-35.030 900 μg) | Sub-Cohort 1.3 (ACI-35.030 1800 μg) | Cohort 1 Placebo | Sub-Cohort 2.1 (JACI-35.054 15 μg) | Sub-Cohort 2.2 (JACI-35.054 60 μg) | Cohort 2 Placebo
Number analyzed (Participants) | 6 | 19 | 6 | 10 | 6 | 6 | 4
mmHg
  Change from baseline to Week 26: number analyzed (Participants) | 1 | 19 | 6 | 8 | 6 | 6 | 4
  Change from baseline to Week 26 | -6.00 (NA) — No Standard Deviation as only 1 participant analyzed | 2.47 (8.790) | 3.67 (5.989) | 2.00 (7.578) | -5.00 (3.795) | -3.17 (7.627) | -8.25 (14.500)
  Change from baseline to Week 50: number analyzed (Participants) | 4 | 18 | 5 | 10 | 6 | 6 | 4
  Change from baseline to Week 50 | -6.75 (2.500) | -0.33 (6.334) | 5.20 (9.203) | -4.20 (6.713) | -1.83 (5.037) | -2.50 (5.167) | -5.00 (8.602)
  Change from baseline to Week 74: number analyzed (Participants) | 4 | 17 | 5 | 10 | 6 | 6 | 4
  Change from baseline to Week 74 | -3.75 (5.377) | 4.76 (8.511) | 1.60 (5.857) | 0.40 (7.412) | -3.33 (6.947) | -3.33 (4.227) | -1.25 (11.325)

5. Primary Outcome: Mean Change From Baseline in Systolic Blood Pressure, ITT Set
Description: At reported visits, systolic blood pressures (mmHg = millimeter of mercury) were measured in sitting position only, after the subject has been sitting down for at least 5 minutes.
  A change from baseline value is defined as the value at post-baseline timepoint minus the baseline value, i.e. post-baseline value - baseline value
Time Frame: as for outcome 4
Population: ITT population (i.e. all randomized subjects who received at least 1 dose of the study drug).
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Sub-Cohort 1.1 (ACI-35.030 300 μg) | Sub-Cohort 1.2 (ACI-35.030 900 μg) | Sub-Cohort 1.3 (ACI-35.030 1800 μg) | Cohort 1 Placebo | Sub-Cohort 2.1 (JACI-35.054 15 μg) | Sub-Cohort 2.2 (JACI-35.054 60 μg) | Cohort 2 Placebo
Number analyzed (Participants) | 6 | 19 | 6 | 10 | 6 | 6 | 4
mmHg
  Change from baseline to Week 26: number analyzed (Participants) | 1 | 19 | 6 | 8 | 6 | 6 | 4
  Change from baseline to Week 26 | -15.00 (NA) — No Standard Deviation as only 1 participant analyzed | 4.11 (16.773) | 9.33 (8.335) | 1.38 (11.388) | -3.17 (9.411) | 3.50 (8.550) | -3.75 (27.861)
  Change from baseline to Week 50: number analyzed (Participants) | 4 | 18 | 5 | 10 | 6 | 6 | 4
  Change from baseline to Week 50 | -5.25 (13.647) | -1.83 (19.242) | 9.20 (9.859) | -2.50 (14.393) | 1.33 (17.535) | 0.67 (5.574) | -1.75 (23.243)
  Change from baseline to Week 74: number analyzed (Participants) | 4 | 17 | 5 | 10 | 6 | 6 | 4
  Change from baseline to Week 74 | -3.75 (15.457) | -1.00 (19.082) | 6.60 (15.421) | -1.60 (21.035) | 0.67 (17.014) | -2.83 (7.195) | 3.75 (27.208)

6. Primary Outcome: Mean Change From Baseline in Heart Rate, ITT Set
Description: At reported visits, heart rates (bpm = beats per minute) were measured in sitting position only, after the subject has been sitting down for at least 5 minutes.
  A change from baseline value is defined as the value at post-baseline timepoint minus the baseline value, i.e. post-baseline value - baseline value
Time Frame: as for outcome 4
Population: ITT population (i.e. all randomized subjects who received at least 1 dose of the study drug).
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Sub-Cohort 1.1 (ACI-35.030 300 μg) | Sub-Cohort 1.2 (ACI-35.030 900 μg) | Sub-Cohort 1.3 (ACI-35.030 1800 μg) | Cohort 1 Placebo | Sub-Cohort 2.1 (JACI-35.054 15 μg) | Sub-Cohort 2.2 (JACI-35.054 60 μg) | Cohort 2 Placebo
Number analyzed (Participants) | 6 | 19 | 6 | 10 | 6 | 6 | 4
bpm
  Change from baseline to Week 26: number analyzed (Participants) | 1 | 19 | 6 | 8 | 6 | 6 | 4
  Change from baseline to Week 26 | -2.00 (NA) — No Standard Deviation as only 1 participant analyzed | -4.11 (9.225) | -1.17 (9.948) | -4.38 (11.649) | -1.83 (7.494) | -0.33 (4.885) | -10.00 (11.888)
  Change from baseline to Week 50: number analyzed (Participants) | 4 | 18 | 5 | 10 | 6 | 6 | 4
  Change from baseline to Week 50 | -5.75 (4.193) | -2.61 (7.935) | -2.80 (7.596) | -0.30 (9.019) | -6.00 (5.762) | -3.00 (6.633) | -7.25 (11.558)
  Change from baseline to Week 74: number analyzed (Participants) | 4 | 17 | 5 | 10 | 6 | 6 | 4
  Change from baseline to Week 74 | 2.25 (6.752) | 1.41 (8.675) | -7.40 (7.232) | 1.90 (13.674) | -6.17 (3.920) | -0.67 (7.967) | -10.25 (14.728)

7. Primary Outcome: Mean Change From Baseline in Body Temperature, ITT Set
Description: At reported visits, body temperatures (°C = degree Celsius) were measured. A change from baseline value is defined as the value at post-baseline timepoint minus the baseline value, i.e. post-baseline value - baseline value
Time Frame: as for outcome 4
Population: ITT population (i.e. all randomized subjects who received at least 1 dose of the study drug).
Measure: Mean (Standard Deviation); unit: °C
Arm/Group | Sub-Cohort 1.1 (ACI-35.030 300 μg) | Sub-Cohort 1.2 (ACI-35.030 900 μg) | Sub-Cohort 1.3 (ACI-35.030 1800 μg) | Cohort 1 Placebo | Sub-Cohort 2.1 (JACI-35.054 15 μg) | Sub-Cohort 2.2 (JACI-35.054 60 μg) | Cohort 2 Placebo
Number analyzed (Participants) | 6 | 19 | 6 | 10 | 6 | 6 | 4
°C
  Change from baseline to Week 26: number analyzed (Participants) | 1 | 19 | 6 | 8 | 6 | 6 | 4
  Change from baseline to Week 26 | -0.40 (NA) — No Standard Deviation as only 1 participant analyzed | 0.02 (0.617) | 0.03 (0.367) | 0.19 (0.360) | 0.12 (0.781) | 0.02 (0.462) | 0.30 (0.497)
  Change from baseline to Week 50: number analyzed (Participants) | 4 | 18 | 5 | 10 | 6 | 6 | 4
  Change from baseline to Week 50 | 0.03 (0.299) | 0.18 (0.451) | -0.04 (0.532) | 0.36 (0.357) | -0.08 (0.880) | -0.47 (0.266) | 0.05 (0.635)
  Change from baseline to Week 74: number analyzed (Participants) | 4 | 17 | 5 | 10 | 6 | 6 | 4
  Change from baseline to Week 74 | 0.08 (0.171) | 0.13 (0.625) | -0.18 (0.383) | 0.29 (0.623) | 0.00 (0.555) | -0.35 (0.367) | 0.15 (0.436)

8. Primary Outcome: Number of Participants Reporting Suicidal Ideation or Behavior Using Columbia-Suicide Severity Rating Scale (C-SSRS), ITT Set
Description: Suicidal ideation or behavior using Columbia-Suicide Severity Rating Scale (C-SSRS) was assessed at Baseline (screening or visit 1 (Week 0)) and at weeks 26, 50 and 74. A set of questions related to suicidal behavior or ideation was directly asked by the rater to the subject.
Time Frame: Endpoint is assessed from baseline (i.e. last non-missing value prior to the first immunization at Visit 1 (Week 0) or Screening) to the last study visit (week 74), at weeks 26, 50 and 74.
Population: ITT population (i.e. all randomized subjects who received at least 1 dose of the study drug).
Measure: Count of Participants; unit: Participants
Arm/Group | Sub-Cohort 1.1 (ACI-35.030 300 μg) | Sub-Cohort 1.2 (ACI-35.030 900 μg) | Sub-Cohort 1.3 (ACI-35.030 1800 μg) | Cohort 1 Placebo | Sub-Cohort 2.1 (JACI-35.054 15 μg) | Sub-Cohort 2.2 (JACI-35.054 60 μg) | Cohort 2 Placebo
Number analyzed (Participants) | 6 | 19 | 6 | 10 | 6 | 6 | 4
Participants
  Suicidal ideation or behavior - Baseline: No | 6 | 19 | 6 | 10 | 6 | 6 | 4
  Suicidal ideation or behavior - Baseline: Yes | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Suicidal ideation or behavior - Week 26: number analyzed (Participants) | 3 | 19 | 6 | 10 | 6 | 6 | 4
  Suicidal ideation or behavior - Week 26: No | 3 | 19 | 6 | 10 | 6 | 6 | 4
  Suicidal ideation or behavior - Week 26: Yes | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Suicidal ideation or behavior - Week 50: number analyzed (Participants) | 4 | 18 | 5 | 10 | 6 | 6 | 4
  Suicidal ideation or behavior - Week 50: No | 4 | 18 | 5 | 10 | 5 | 6 | 4
  Suicidal ideation or behavior - Week 50: Yes | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Suicidal ideation or behavior - Week 74: number analyzed (Participants) | 4 | 17 | 5 | 10 | 6 | 6 | 4
  Suicidal ideation or behavior - Week 74: No | 4 | 17 | 5 | 10 | 6 | 6 | 4
  Suicidal ideation or behavior - Week 74: Yes | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Primary Outcome: Number of Participants With Abnormal MRI Results, ITT Set
Description: Brain MRI scans were conducted according to the schedule of assessments, i.e. at Baseline (screening) and at weeks 10, 26, 50, 74 and examined for evidence of brain pathology. Normal, abnormal not clinically significant (NCS) and abnormal clinically significant (CS) results as interpreted by the clinical site are reported.
Time Frame: Endpoint is assessed from baseline (screening) to the last study visit (week 74), at weeks 10, 26, 50 and 74.
Population: ITT population (i.e. all randomized subjects who received at least 1 dose of the study drug).
Measure: Count of Participants; unit: Participants
Arm/Group | Sub-Cohort 1.1 (ACI-35.030 300 μg) | Sub-Cohort 1.2 (ACI-35.030 900 μg) | Sub-Cohort 1.3 (ACI-35.030 1800 μg) | Cohort 1 Placebo | Sub-Cohort 2.1 (JACI-35.054 15 μg) | Sub-Cohort 2.2 (JACI-35.054 60 μg) | Cohort 2 Placebo
Number analyzed (Participants) | 6 | 19 | 6 | 10 | 6 | 6 | 4
Participants
  Baseline: Normal | 5 | 17 | 6 | 10 | 5 | 6 | 4
  Baseline: Abnormal NCS | 1 | 2 | 0 | 0 | 1 | 0 | 0
  Baseline: Abnormal CS | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Baseline: Not evaluable | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 10: Normal | 6 | 16 | 6 | 10 | 6 | 6 | 4
  Week 10: Abnormal NCS | 0 | 2 | 0 | 0 | 0 | 0 | 0
  Week 10: Abnormal CS | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 10: Not evaluable | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Week 26: number analyzed (Participants) | 1 | 19 | 6 | 8 | 6 | 6 | 4
  Week 26: Normal | 1 | 17 | 6 | 7 | 6 | 6 | 4
  Week 26: Abnormal NCS | 0 | 2 | 0 | 0 | 0 | 0 | 0
  Week 26: Abnormal CS | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 26: Not evaluable | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Week 50: number analyzed (Participants) | 4 | 18 | 5 | 10 | 6 | 6 | 4
  Week 50: Normal | 4 | 17 | 5 | 10 | 6 | 5 | 4
  Week 50: Abnormal NCS | 0 | 1 | 0 | 0 | 0 | 1 | 0
  Week 50: Abnormal CS | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 50: Not evaluable | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 74: number analyzed (Participants) | 3 | 17 | 5 | 10 | 6 | 6 | 4
  Week 74: Normal | 3 | 15 | 5 | 10 | 6 | 4 | 3
  Week 74: Abnormal NCS | 0 | 2 | 0 | 0 | 0 | 2 | 1
  Week 74: Abnormal CS | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 74: Not evaluable | 0 | 0 | 0 | 0 | 0 | 0 | 0

10. Primary Outcome: Anti-pTau IgG Antibody Response in Serum - Antibody Titers, ITT Set
Description: At all visits, blood was collected for the determination of the immune response in serum. Anti-phosphorylated Tau (pTau) IgG titers were measured by Meso Scale Discovery (MSD). For each visit, the geometric means (AU/mL) and 95% Confidence Interval (CI) is given.
Time Frame: Endpoint is assessed from baseline (i.e. mean of the titers measured at the screening and visit 1 before the first study drug administration) to the last study visit (week 74), at weeks 0, 2, 8, 10, 24, 26, 36, 48, 50, 67 and 74.
Population: ITT population (i.e. all randomized subjects who received at least 1 dose of the study drug).
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | Sub-Cohort 1.1 (ACI-35.030 300 μg) | Sub-Cohort 1.2 (ACI-35.030 900 μg) | Sub-Cohort 1.3 (ACI-35.030 1800 μg) | Cohort 1 Placebo | Sub-Cohort 2.1 (JACI-35.054 15 μg) | Sub-Cohort 2.2 (JACI-35.054 60 μg) | Cohort 2 Placebo
Number analyzed (Participants) | 6 | 19 | 6 | 10 | 6 | 6 | 4
AU/mL
  Baseline | 2048.4 [1155.4 to 3631.6] | 994.6 [688.7 to 1436.5] | 676.2 [476.0 to 960.6] | 802.4 [713.5 to 902.2] | 913.9 [619.4 to 1348.4] | 1073.3 [808.9 to 1424.1] | 981.7 [711.2 to 1354.9]
  Week 2 | 80292.0 [37517.3 to 171835.3] | 158154.6 [86332.2 to 289728.2] | 187980.6 [99157.0 to 356371.2] | 811.0 [714.5 to 920.5] | 1403.8 [1065.4 to 1849.6] | 5286.1 [1053.3 to 26530.2] | 895.4 [598.7 to 1339.2]
  Week 8 | 49360.9 [19121.1 to 127424.7] | 92181.7 [56336.9 to 150833.0] | 66035.9 [37536.0 to 116174.9] | 768.6 [684.5 to 863.1] | 3054.4 [1875.2 to 4975.1] | 6928.5 [2386.1 to 20118.9] | 971.5 [668.5 to 1412.0]
  Week 10 | 110984.4 [31648.6 to 389197.3] | 182111.4 [113522.2 to 292141.7] | 135520.1 [71679.7 to 256219.1] | 749.7 [652.5 to 861.4] | 105042.6 [39205.0 to 281442.5] | 82513.4 [34350.2 to 198207.6] | 969.2 [671.7 to 1398.6]
  Week 24: number analyzed (Participants) | 1 | 19 | 6 | 8 | 6 | 6 | 4
  Week 24 | 6900.0 [NA to NA] — No Confidence Interval as only 1 participant analyzed | 32248.7 [19704.9 to 52777.7] | 19853.3 [10110.8 to 38983.4] | 1056.1 [860.3 to 1296.6] | 27519.3 [11321.5 to 66891.5] | 27030.2 [11647.9 to 62726.3] | 789.4 [524.8 to 1187.3]
  Week 26: number analyzed (Participants) | 1 | 18 | 6 | 8 | 6 | 6 | 4
  Week 26 | 21800.0 [NA to NA] — No Confidence Interval as only 1 participant analyzed | 71385.3 [43249.5 to 117824.7] | 60104.8 [26253.5 to 137603.9] | 1136.8 [913.4 to 1414.8] | 329361.3 [136886.4 to 792473.2] | 123787.7 [85919.6 to 178345.7] | 919.5 [646.4 to 1308.0]
  Week 36: number analyzed (Participants) | 6 | 18 | 6 | 10 | 6 | 6 | 4
  Week 36 | 8207.3 [3347.2 to 20124.4] | 30141.2 [17057.1 to 53261.7] | 19810.7 [9322.3 to 42099.2] | 571.6 [373.6 to 874.5] | 127585.6 [64839.7 to 251051.1] | 58190.1 [43600.4 to 77661.9] | 1245.1 [728.7 to 2127.6]
  Week 48: number analyzed (Participants) | 4 | 18 | 5 | 10 | 6 | 5 | 4
  Week 48 | 5408.4 [2873.1 to 10181.1] | 17533.0 [9904.6 to 31036.7] | 10848.2 [4285.7 to 27459.9] | 676.2 [523.4 to 873.7] | 56549.1 [28051.0 to 113999.4] | 25968.2 [18637.2 to 36182.9] | 1137.1 [599.1 to 2158.2]
  Week 50: number analyzed (Participants) | 4 | 18 | 5 | 10 | 6 | 6 | 4
  Week 50 | 86662.7 [22301.9 to 336760.7] | 54164.6 [28561.9 to 102717.6] | 63735.9 [38946.7 to 104303.4] | 617.0 [464.4 to 819.7] | 408403.6 [273922.2 to 608908.1] | 137934.8 [61731.7 to 308205.1] | 1311.8 [750.6 to 2292.6]
  Week 67: number analyzed (Participants) | 4 | 17 | 5 | 10 | 6 | 6 | 4
  Week 67 | 14623.7 [7565.4 to 28267.4] | 17464.2 [8728.8 to 34941.7] | 10128.3 [5232.7 to 19604.1] | 714.1 [555.9 to 917.2] | 144349.8 [92815.9 to 224496.7] | 47764.4 [20377.3 to 111959.5] | 681.2 [451.3 to 1028.0]
  Week 74: number analyzed (Participants) | 4 | 17 | 5 | 10 | 6 | 6 | 4
  Week 74 | 10527.5 [6075.0 to 18243.5] | 15301.0 [7889.7 to 29673.9] | 8565.4 [3914.9 to 18740.2] | 719.1 [577.5 to 895.5] | 107038.5 [63784.9 to 179623.2] | 31817.4 [11556.3 to 87601.2] | 682.9 [468.2 to 995.9]

11. Primary Outcome: Anti-ePHF IgG Antibody Response in Serum - Antibody Titers, ITT Set
Description: At all visits, blood was collected for the determination of the immune response in serum. Anti-enriched paired helical filaments (ePHF) IgG titers were measured by Meso Scale Discovery (MSD). For each visit, the geometric means (AU/mL) and 95% Confidence Interval (CI) is given.
Time Frame: as for outcome 10
Population: ITT population (i.e. all randomized subjects who received at least 1 dose of the study drug)
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | Sub-Cohort 1.1 (ACI-35.030 300 μg) | Sub-Cohort 1.2 (ACI-35.030 900 μg) | Sub-Cohort 1.3 (ACI-35.030 1800 μg) | Cohort 1 Placebo | Sub-Cohort 2.1 (JACI-35.054 15 μg) | Sub-Cohort 2.2 (JACI-35.054 60 μg) | Cohort 2 Placebo
Number analyzed (Participants) | 6 | 19 | 6 | 10 | 6 | 6 | 4
AU/mL
  Baseline | 1553.4 [1116.9 to 2160.5] | 2515.4 [1449.4 to 4365.5] | 1691.8 [862.3 to 3319.3] | 2006.5 [1120.3 to 3593.7] | 2659.9 [1508.2 to 4691.1] | 2027.6 [1551.2 to 2650.4] | 2754.4 [1696.8 to 4471.2]
  Week 2 | 4147.0 [1790.9 to 9602.7] | 8245.3 [5162.3 to 13169.5] | 4132.5 [2007.6 to 8506.3] | 2270.6 [1276.5 to 4038.9] | 2419.2 [1263.7 to 4631.6] | 2128.4 [1371.1 to 3303.9] | 2680.9 [1514.7 to 4745.2]
  Week 8 | 4281.7 [2522.5 to 7267.8] | 7928.5 [5215.6 to 12052.4] | 3973.2 [2439.9 to 6469.9] | 1992.7 [1095.7 to 3624.2] | 2904.3 [1461.7 to 5770.6] | 2270.4 [1289.0 to 3999.3] | 2682.9 [1663.9 to 4326.0]
  Week 10 | 9371.5 [3398.3 to 25843.8] | 17848.1 [11623.1 to 27406.9] | 9317.6 [5404.3 to 16064.5] | 2099.3 [1172.8 to 3757.7] | 17874.8 [8298.9 to 38500.1] | 13086.9 [6317.8 to 27108.8] | 2497.6 [1493.9 to 4175.7]
  Week 24: number analyzed (Participants) | 1 | 19 | 6 | 8 | 6 | 6 | 4
  Week 24 | 2770.0 [NA to NA] — No Confidence Interval as only 1 participant analyzed | 9446.6 [6001.8 to 14868.6] | 6424.4 [2758.4 to 14962.3] | 2381.2 [1081.9 to 5241.0] | 6235.7 [3717.7 to 10459.3] | 5275.9 [3016.0 to 9228.9] | 2128.9 [923.8 to 4906.4]
  Week 26: number analyzed (Participants) | 1 | 18 | 6 | 8 | 6 | 6 | 4
  Week 26 | 3890.0 [NA to NA] — No Confidence Interval as only 1 participant analyzed | 13142.7 [8034.0 to 21499.9] | 8779.5 [4383.4 to 17584.7] | 2488.8 [1181.0 to 5244.9] | 32099.1 [10656.3 to 96688.8] | 17640.8 [12002.0 to 25928.7] | 2174.3 [918.7 to 5146.0]
  Week 36: number analyzed (Participants) | 6 | 18 | 6 | 10 | 6 | 6 | 4
  Week 36 | 2709.4 [2188.5 to 3354.3] | 12713.9 [7440.1 to 21726.0] | 6886.6 [2758.6 to 17191.7] | 2358.4 [1297.9 to 4285.5] | 14491.7 [6314.7 to 33257.6] | 10543.9 [7864.9 to 14135.6] | 2273.8 [1091.3 to 4737.7]
  Week 48: number analyzed (Participants) | 4 | 18 | 5 | 10 | 6 | 5 | 4
  Week 48 | 2287.7 [1733.1 to 3019.9] | 9108.4 [5469.1 to 15169.4] | 5886.6 [2446.7 to 14162.3] | 2254.2 [1218.0 to 4171.7] | 7237.2 [3437.4 to 15237.7] | 6321.2 [4670.3 to 8555.7] | 2213.5 [969.2 to 5055.1]
  Week 50: number analyzed (Participants) | 4 | 18 | 5 | 10 | 6 | 6 | 4
  Week 50 | 7472.5 [3323.2 to 16802.6] | 13280.3 [7620.5 to 23143.7] | 8536.0 [4170.1 to 17472.6] | 2340.1 [1268.6 to 4317.0] | 30248.2 [12315.3 to 74294.5] | 25491.5 [10441.9 to 62231.3] | 2436.9 [1199.6 to 4950.6]
  Week 67: number analyzed (Participants) | 4 | 17 | 5 | 10 | 6 | 6 | 4
  Week 67 | 3219.8 [2578.6 to 4020.4] | 8944.8 [5974.4 to 13392.0] | 6180.6 [2623.0 to 14563.1] | 2080.4 [1122.4 to 3856.0] | 13077.0 [7162.9 to 23874.1] | 10082.0 [4602.9 to 22083.5] | 2295.7 [1480.2 to 3560.6]
  Week 74: number analyzed (Participants) | 4 | 17 | 5 | 10 | 6 | 6 | 4
  Week 74 | 2791.9 [2285.3 to 3410.8] | 8993.0 [5314.7 to 15216.9] | 5383.9 [2349.5 to 12337.4] | 2126.0 [1168.7 to 3867.5] | 10835.5 [5870.1 to 20000.8] | 6788.7 [3017.2 to 15274.3] | 2178.8 [1549.6 to 3063.5]

12. Secondary Outcome: Anti-Tau IgG Antibody Response in Serum - Antibody Titers, ITT Set
Description: At all visits, blood was collected for the determination of the immune response in serum. Anti-Tau IgG titers were measured by Meso Scale Discovery (MSD). For each visit, the geometric means (AU/mL) and 95% Confidence Interval (CI) is given.
Time Frame: as for outcome 10
Population: ITT population (i.e. all randomized subjects who received at least 1 dose of the study drug)
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | Sub-Cohort 1.1 (ACI-35.030 300 μg) | Sub-Cohort 1.2 (ACI-35.030 900 μg) | Sub-Cohort 1.3 (ACI-35.030 1800 μg) | Cohort 1 Placebo | Sub-Cohort 2.1 (JACI-35.054 15 μg) | Sub-Cohort 2.2 (JACI-35.054 60 μg) | Cohort 2 Placebo
Number analyzed (Participants) | 6 | 19 | 6 | 10 | 6 | 6 | 4
AU/mL
  Baseline | 374.7 [287.3 to 488.8] | 357.1 [238.3 to 535.2] | 355.4 [125.2 to 1008.8] | 251.7 [198.1 to 319.7] | 223.0 [135.4 to 367.5] | 394.1 [290.2 to 535.3] | 261.0 [144.2 to 472.4]
  Week 2 | 2609.5 [1098.9 to 6196.6] | 8753.9 [3767.6 to 20339.8] | 6549.6 [1614.8 to 26564.8] | 230.4 [186.1 to 285.1] | 744.5 [390.0 to 1421.1] | 2657.0 [524.4 to 13461.1] | 233.7 [118.9 to 459.4]
  Week 8 | 1065.0 [512.3 to 2213.9] | 3631.9 [1709.8 to 7714.8] | 2000.8 [704.1 to 5685.1] | 243.1 [192.6 to 306.7] | 2564.1 [1753.4 to 3749.5] | 4349.6 [1372.9 to 13780.8] | 253.3 [132.3 to 484.9]
  Week 10 | 1508.6 [649.3 to 3505.4] | 4217.5 [2120.6 to 8387.6] | 2921.6 [1391.6 to 6133.8] | 242.5 [208.3 to 282.4] | 84688.8 [36848.8 to 194638.7] | 46411.7 [23609.7 to 91235.4] | 262.8 [106.9 to 646.4]
  Week 24: number analyzed (Participants) | 1 | 19 | 6 | 8 | 6 | 6 | 4
  Week 24 | 578.0 [NA to NA] — No Confidence Interval as only 1 participant analyzed | 1124.8 [647.0 to 1955.5] | 851.6 [364.5 to 1989.6] | 343.3 [285.9 to 412.2] | 16444.7 [6570.8 to 41155.8] | 19762.7 [8882.8 to 43968.6] | 236.2 [130.0 to 429.2]
  Week 26: number analyzed (Participants) | 1 | 18 | 6 | 8 | 6 | 6 | 4
  Week 26 | 798.0 [NA to NA] — No Confidence Interval as only 1 participant analyzed | 1375.2 [980.6 to 1928.6] | 1859.0 [867.8 to 3982.4] | 339.5 [262.9 to 438.2] | 162241.1 [72817.9 to 361479.1] | 74795.1 [40734.0 to 137337.3] | 237.9 [139.4 to 406.1]
  Week 36: number analyzed (Participants) | 6 | 18 | 6 | 10 | 6 | 6 | 4
  Week 36 | 523.3 [358.4 to 764.1] | 828.6 [458.0 to 1499.1] | 806.3 [306.5 to 2121.3] | 240.6 [180.5 to 320.6] | 59209.8 [35862.2 to 97757.4] | 31504.2 [19187.4 to 51727.4] | 310.1 [170.6 to 563.7]
  Week 48: number analyzed (Participants) | 4 | 18 | 5 | 10 | 6 | 5 | 4
  Week 48 | 416.0 [279.6 to 618.9] | 635.2 [354.9 to 1136.9] | 417.1 [212.1 to 820.1] | 243.1 [181.6 to 325.4] | 25681.2 [14983.1 to 44017.8] | 13486.3 [7865.4 to 23124.1] | 282.8 [153.1 to 522.4]
  Week 50: number analyzed (Participants) | 4 | 18 | 5 | 10 | 6 | 6 | 4
  Week 50 | 1023.0 [594.5 to 1760.3] | 1092.4 [595.6 to 2003.5] | 1132.9 [472.2 to 2718.2] | 231.8 [172.2 to 312.0] | 197833.5 [123950.4 to 315756.0] | 70122.6 [32136.3 to 153009.8] | 286.5 [157.2 to 522.1]
  Week 67: number analyzed (Participants) | 4 | 17 | 5 | 10 | 6 | 6 | 4
  Week 67 | 450.1 [342.4 to 591.7] | 551.2 [321.7 to 944.6] | 570.6 [329.0 to 989.6] | 269.6 [205.4 to 353.8] | 69607.0 [43695.0 to 110885.3] | 32158.7 [12000.4 to 86178.7] | 282.6 [213.5 to 374.0]
  Week 74: number analyzed (Participants) | 4 | 17 | 5 | 10 | 6 | 6 | 4
  Week 74 | 439.4 [366.2 to 527.3] | 590.0 [327.6 to 1062.4] | 571.9 [334.2 to 978.6] | 253.3 [172.3 to 372.5] | 51718.4 [30576.2 to 87479.7] | 21920.5 [7062.2 to 68039.9] | 267.4 [156.3 to 457.3]

13. Secondary Outcome: Anti-pTau IgM Antibody Response in Serum - Antibody Titers, ITT Set
Description: At all visits, blood was collected for the determination of the immune response in serum. Anti-phosphorylated Tau (pTau) IgM titers were measured by enzyme-linked immunosorbent assay (ELISA). For each visit, the geometric means (AU/mL) and 95% Confidence Interval (CI) is given.
Time Frame: as for outcome 10
Population: ITT population (i.e. all randomized subjects who received at least 1 dose of the study drug).
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | Sub-Cohort 1.1 (ACI-35.030 300 μg) | Sub-Cohort 1.2 (ACI-35.030 900 μg) | Sub-Cohort 1.3 (ACI-35.030 1800 μg) | Cohort 1 Placebo | Sub-Cohort 2.1 (JACI-35.054 15 μg) | Sub-Cohort 2.2 (JACI-35.054 60 μg) | Cohort 2 Placebo
Number analyzed (Participants) | 6 | 19 | 6 | 10 | 6 | 6 | 4
AU/mL
  Baseline | 355.3 [162.5 to 777.0] | 154.8 [113.9 to 210.4] | 368.6 [247.9 to 547.9] | 297.5 [166.8 to 530.6] | 337.3 [190.5 to 597.4] | 147.1 [50.2 to 431.4] | 248.5 [100.0 to 617.5]
  Week 2 | 25951.9 [11858.8 to 56793.5] | 15563.7 [10500.7 to 23067.8] | 20464.3 [6475.2 to 64676.0] | 297.5 [167.9 to 527.4] | 494.9 [236.3 to 1036.2] | 327.4 [100.9 to 1062.4] | 237.2 [76.6 to 734.5]
  Week 8 | 3666.8 [1795.4 to 7488.6] | 3439.4 [2477.0 to 4775.7] | 4936.6 [1625.2 to 14994.8] | 274.9 [158.5 to 476.8] | 476.8 [241.0 to 943.4] | 276.8 [108.5 to 706.1] | 217.4 [76.7 to 615.9]
  Week 10 | 4436.9 [2723.2 to 7229.1] | 4792.5 [3376.5 to 6802.3] | 7672.5 [3433.5 to 17144.9] | 288.5 [165.5 to 503.0] | 564.7 [266.4 to 1197.1] | 349.6 [139.2 to 877.8] | 225.5 [74.3 to 684.3]
  Week 24: number analyzed (Participants) | 1 | 19 | 6 | 8 | 6 | 6 | 4
  Week 24 | 696.0 [NA to NA] — No Confidence Interval as only 1 participant analyzed | 1967.4 [1598.0 to 2422.3] | 2758.4 [1380.1 to 5513.0] | 345.0 [158.5 to 750.9] | 473.9 [215.5 to 1042.1] | 202.6 [118.6 to 346.0] | 183.3 [66.6 to 504.3]
  Week 26: number analyzed (Participants) | 1 | 18 | 6 | 8 | 6 | 6 | 4
  Week 26 | 2830.0 [NA to NA] — No Confidence Interval as only 1 participant analyzed | 5137.1 [3815.8 to 6916.0] | 7950.1 [3857.6 to 16384.4] | 334.8 [154.6 to 725.2] | 483.3 [213.7 to 1093.0] | 153.5 [69.1 to 341.1] | 181.8 [64.9 to 509.6]
  Week 36: number analyzed (Participants) | 6 | 18 | 6 | 10 | 6 | 6 | 4
  Week 36 | 806.2 [394.4 to 1647.9] | 2958.8 [2148.6 to 4074.6] | 2906.2 [1516.6 to 5569.2] | 308.2 [168.4 to 564.0] | 356.1 [204.2 to 621.2] | 329.0 [143.4 to 754.5] | 265.4 [83.0 to 848.1]
  Week 48: number analyzed (Participants) | 4 | 18 | 5 | 10 | 6 | 5 | 4
  Week 48 | 802.9 [383.6 to 1680.4] | 1789.3 [1318.7 to 2428.0] | 2362.7 [1131.0 to 4935.4] | 310.9 [173.0 to 558.5] | 368.6 [199.9 to 679.7] | 297.6 [91.5 to 967.3] | 278.1 [84.2 to 919.0]
  Week 50: number analyzed (Participants) | 4 | 18 | 5 | 10 | 6 | 6 | 4
  Week 50 | 4714.6 [1996.9 to 11131.2] | 5214.3 [3348.3 to 8120.3] | 8509.3 [3839.7 to 18857.4] | 318.9 [174.9 to 581.1] | 360.5 [215.5 to 603.1] | 248.8 [92.0 to 672.8] | 275.0 [84.3 to 897.1]
  Week 67: number analyzed (Participants) | 4 | 17 | 5 | 10 | 6 | 6 | 4
  Week 67 | 1858.5 [879.0 to 3929.7] | 1898.6 [1275.1 to 2827.0] | 4539.9 [2155.0 to 9564.3] | 431.9 [233.9 to 797.3] | 393.7 [199.1 to 778.7] | 240.5 [73.6 to 785.3] | 186.7 [57.9 to 602.1]
  Week 74: number analyzed (Participants) | 4 | 17 | 5 | 10 | 6 | 6 | 4
  Week 74 | 1785.9 [801.8 to 3977.8] | 1509.7 [1063.2 to 2143.7] | 3880.2 [1741.4 to 8645.9] | 343.0 [191.9 to 613.3] | 449.9 [248.2 to 815.4] | 252.9 [75.6 to 845.9] | 348.0 [79.0 to 1533.3]

14. Secondary Outcome: Anti-Tau IgM Antibody Response in Serum - Antibody Titers, ITT Set
Description: At all visits, blood was collected for the determination of the immune response in serum. Anti-Tau IgM titers were measured by enzyme-linked immunosorbent assay (ELISA). For each visit, the geometric means (AU/mL) and 95% Confidence Interval (CI) is given.
Time Frame: as for outcome 10
Population: ITT population (i.e. all randomized subjects who received at least 1 dose of the study drug).
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | Sub-Cohort 1.1 (ACI-35.030 300 μg) | Sub-Cohort 1.2 (ACI-35.030 900 μg) | Sub-Cohort 1.3 (ACI-35.030 1800 μg) | Cohort 1 Placebo | Sub-Cohort 2.1 (JACI-35.054 15 μg) | Sub-Cohort 2.2 (JACI-35.054 60 μg) | Cohort 2 Placebo
Number analyzed (Participants) | 6 | 19 | 6 | 10 | 6 | 6 | 4
AU/mL
  Baseline | 153.0 [69.6 to 336.2] | 93.1 [66.8 to 129.6] | 124.4 [64.0 to 241.9] | 108.1 [73.4 to 159.2] | 93.7 [42.9 to 204.8] | 94.6 [36.6 to 244.7] | 119.3 [44.3 to 321.4]
  Week 2 | 460.7 [185.3 to 1145.2] | 449.8 [222.5 to 909.6] | 737.8 [121.6 to 4478.3] | 105.4 [70.0 to 158.6] | 146.1 [56.5 to 378.0] | 139.6 [48.2 to 404.2] | 129.9 [43.7 to 386.3]
  Week 8 | 228.3 [107.3 to 485.6] | 209.6 [127.3 to 345.0] | 333.4 [72.0 to 1543.1] | 98.2 [67.3 to 143.5] | 116.8 [53.7 to 253.8] | 101.3 [38.4 to 267.2] | 116.5 [44.1 to 307.8]
  Week 10 | 220.8 [135.4 to 360.0] | 209.5 [133.8 to 328.0] | 409.5 [127.0 to 1320.6] | 101.3 [68.9 to 148.8] | 119.2 [54.3 to 261.3] | 123.2 [46.5 to 326.2] | 117.4 [43.6 to 316.0]
  Week 24: number analyzed (Participants) | 1 | 18 | 6 | 8 | 6 | 6 | 4
  Week 24 | 231.0 [NA to NA] — No Confidence Interval as only 1 participant analyzed | 134.2 [98.3 to 183.0] | 181.2 [75.1 to 437.3] | 90.2 [63.3 to 128.5] | 100.8 [51.3 to 198.2] | 102.3 [46.0 to 227.6] | 104.1 [40.1 to 270.4]
  Week 26: number analyzed (Participants) | 1 | 18 | 6 | 8 | 6 | 6 | 4
  Week 26 | 256.0 [NA to NA] — No Confidence Interval as only 1 participant analyzed | 198.8 [158.9 to 248.7] | 286.2 [136.2 to 601.6] | 87.2 [57.4 to 132.5] | 107.9 [53.3 to 218.8] | 105.9 [48.0 to 233.8] | 103.3 [40.8 to 261.4]
  Week 36: number analyzed (Participants) | 6 | 18 | 6 | 10 | 6 | 6 | 4
  Week 36 | 95.2 [51.2 to 177.0] | 264.6 [198.1 to 353.3] | 476.7 [282.4 to 804.7] | 107.7 [61.5 to 188.7] | 101.1 [51.4 to 198.9] | 100.1 [37.2 to 268.9] | 147.4 [58.1 to 373.9]
  Week 48: number analyzed (Participants) | 4 | 18 | 5 | 10 | 6 | 5 | 4
  Week 48 | 111.6 [43.0 to 289.6] | 232.9 [178.6 to 303.8] | 468.3 [191.5 to 1145.1] | 120.9 [70.7 to 206.9] | 125.8 [67.3 to 235.1] | 133.4 [45.6 to 390.7] | 162.6 [62.6 to 422.4]
  Week 50: number analyzed (Participants) | 4 | 18 | 5 | 10 | 6 | 6 | 4
  Week 50 | 171.9 [74.8 to 395.0] | 349.2 [270.4 to 450.9] | 507.4 [227.5 to 1131.9] | 108.3 [61.3 to 191.2] | 102.4 [52.2 to 201.0] | 110.1 [44.3 to 274.1] | 164.9 [65.0 to 418.2]
  Week 67: number analyzed (Participants) | 4 | 17 | 5 | 10 | 6 | 6 | 4
  Week 67 | 147.8 [61.5 to 355.0] | 202.7 [142.6 to 288.0] | 342.5 [116.4 to 1007.7] | 109.7 [70.9 to 169.6] | 93.1 [43.0 to 201.5] | 130.9 [49.2 to 348.2] | 144.9 [54.7 to 384.0]
  Week 74: number analyzed (Participants) | 4 | 17 | 5 | 10 | 6 | 6 | 4
  Week 74 | 144.1 [43.4 to 478.7] | 169.1 [121.8 to 234.6] | 329.9 [111.9 to 972.3] | 128.2 [90.0 to 182.6] | 108.4 [51.4 to 228.6] | 130.6 [49.2 to 346.3] | 161.8 [58.5 to 447.2]

15. Other Pre Specified Outcome: Change From Baseline of Functional Performance Using CDR-SB Scale
Description: CDR-SB means Clinical Dementia Rating - Sum of Boxes. The score ranges from 0 to 18. A higher score indicates a worse outcome.
Time Frame: from baseline up to week 74
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Change From Baseline of Cognitive Performance Using RBANS Scale
Description: RBANS means Repeatable Battery for the Assessment of Neuropsychological Status. The total scale index score ranges from 40 to 160. A higher score indicates a better outcome.
Time Frame: from baseline up to week 74
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Change From Baseline of Behavior Using NPI Scale
Description: NPI means Neuropsychiatric Inventory. The score ranges from 0 to 144. A higher score indicates a worse outcome.
Time Frame: from baseline up to week 74
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: The safety reporting period covering any Adverse Events which were treatment-emergent is the interval between the first dosing (Visit 1, Week 0) and the last safety follow-up visit (Visit 11, Week 74); up to 74 weeks.
Description: Determination of Adverse Events was based on:
  * the signs or symptoms detected during the physical examination of the subject and on clinical assessments (e.g. laboratory values, MRI results etc.)
  * the interview of the subject and their caregiver
Arm/Group | Sub-Cohort 1.1 (ACI-35.030 300 μg) | Sub-Cohort 1.2 (ACI-35.030 900 μg) | Sub-Cohort 1.3 (ACI-35.030 1800 μg) | Cohort 1 Placebo | Sub-Cohort 2.1 (JACI-35.054 15 μg) | Sub-Cohort 2.2 (JACI-35.054 60 μg) | Cohort 2 Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/19 | 0/6 | 0/10 | 0/6 | 0/6 | 0/4
Serious Adverse Events (participants affected / at risk) | 2/6 | 2/19 | 2/6 | 0/10 | 0/6 | 0/6 | 1/4
Other Adverse Events (participants affected / at risk) | 6/6 | 17/19 | 6/6 | 8/10 | 6/6 | 6/6 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sub-Cohort 1.1 (ACI-35.030 300 μg) (N=6) | Sub-Cohort 1.2 (ACI-35.030 900 μg) (N=19) | Sub-Cohort 1.3 (ACI-35.030 1800 μg) (N=6) | Cohort 1 Placebo (N=10) | Sub-Cohort 2.1 (JACI-35.054 15 μg) (N=6) | Sub-Cohort 2.2 (JACI-35.054 60 μg) (N=6) | Cohort 2 Placebo (N=4)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic fever with renal syndrome (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site rash (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aneurysm thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral artery aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sub-Cohort 1.1 (ACI-35.030 300 μg) (N=6) | Sub-Cohort 1.2 (ACI-35.030 900 μg) (N=19) | Sub-Cohort 1.3 (ACI-35.030 1800 μg) (N=6) | Cohort 1 Placebo (N=10) | Sub-Cohort 2.1 (JACI-35.054 15 μg) (N=6) | Sub-Cohort 2.2 (JACI-35.054 60 μg) (N=6) | Cohort 2 Placebo (N=4)
Injection site reaction (General disorders) | 2 (2) | 14 (31) | 6 (9) | 0 (0) | 1 (2) | 2 (3) | 0 (0)
Fatigue (General disorders) | 0 (0) | 4 (4) | 1 (2) | 2 (4) | 0 (0) | 1 (2) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 7 (8) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 3 (4) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (3)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronavirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Otitis media chronic (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 4 (7) | 3 (7) | 0 (0) | 2 (7) | 1 (3) | 1 (2)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Balance disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral microhaemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dementia Alzheimer's type (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Head discomfort (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Postural tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural headache (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stress fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nail injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Salivary gland calculus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (4) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Depressive symptom (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Behaviour disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nightmare (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Blood pressure decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Blood sodium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood iron decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Deafness unilateral (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gaze palsy (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swelling of eyelid (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Epiretinal membrane (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral artery aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
* The study was not powered to detect differences between the active and placebo treatments for exploratory endpoints (e.g., fluid biomarkers and cognition/clinical efficacy outcomes).
* The sub-cohort 1.1 (ACI-35.030 300 μg / placebo) was significantly impacted by the COVID-19 pandemic due to local travel restriction in Finland. Seven out of 8 subjects (5 active and 2 placebo) in this sub-cohort missed 1 study treatment administration.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication shall not be made by PIs before a first multi-site publication by Sponsor. If no multi-site publication is made within 18 months after study completion, PIs can publish under conditions: Prior any publication submission, PI shall send Sponsor any information to be disclosed and Sponsor have 60 days from receipt to review and comment. PI shall remove any Confidential Information and upon Sponsor request further delay publication for up to 120 days to protect Sponsor interests.

DOCUMENTS (2):
  • Study Protocol (2021-10-22): https://cdn.clinicaltrials.gov/large-docs/31/NCT04445831/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-05): https://cdn.clinicaltrials.gov/large-docs/31/NCT04445831/SAP_001.pdf